CLINICAL TRIAL: NCT07099872
Title: Efficacy of a Novel Exercise + Overdressing Protocol to Induce Heat Acclimation in Temperate Environments (Chronic XO-Study)
Brief Title: Chronic Exercise With Overdressing
Acronym: Chronic-XO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-26
Record Dates: First submitted 2025-06-26; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Heat Acclimation and Thermotolerance
Keywords: Heat Acclimation; Heat Stress Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with Overdressing (Experimental): 5 days of standardized exercise with overdressing
  Interventions: Other: Overdressing
- Exercise (Active Comparator): 5 days of standardized exercise wearing PT clothing
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Wear normal attire (shorts/t-shirt) during exercise sessions in a gym-like environment.
  Arms: Exercise
Other: Overdressing — Wear standardized overdressing ensemble during exercise sessions in a gym-like environment.
  Arms: Exercise with Overdressing

SUMMARY:
The purpose of this study is to determine if five training sessions of exercise with overdressing can induce heat acclimation.

DETAILED DESCRIPTION:
Twelve healthy and fit adults will complete 90 min of exercise (6.0 mph run for 30 min followed by 3.5 mph walk for 60 min) on five occasions at room temperature (~20 °C, 50% RH, 1 mph air velocity). Participants will be randomized into either the exercise with overdressing or exercise wearing standard physical training (PT) clothing group and complete the study in a crossover manner. Heat acclimation induction will be assessed using standardized heat stress tests (HSTs) performed before and after five training sessions. After the final HST has occurred, participants will complete a minimum 4-week washout and then return to repeat the identical protocol in the opposite configuration (overdressing vs. PT clothing). The investigators hypothesize that, compared to 5 days of exercise in PT clothing, 5 days of exercise with overdressing will lower end-exercise core temperature during standardized HSTs.

ELIGIBILITY:
Inclusion Criteria:

* Females must be premenopausal.
* Body mass index 18.5-33.0 kg m-2.
* In good health as determined by the Office of Medical Support & Oversight (OMSO) General Medical Clearance.
* Performs aerobic exercise at least 2 times per week and capable of running 2 miles in under 17:00 (8:30 minute mile pace).
* Willing to abstain from exercise and alcoholic beverages for 24 hrs before each study visit.
* Willing to abstain from caffeine for 12 hrs prior to all study visits.
* Willing to abstain from food for 2 hrs prior to all study visits.
* Willing to abstain from nicotine/tobacco for at least 8 hrs prior to all study visits.
* Have supervisor approval if permanent party military or a federal employee at U.S. Army Natick Soldier System Center.

Exclusion Criteria:

* Frequent hot bath or sauna users (e.g., more than three times a week for the past month).
* Females who are pregnant or planning to become pregnant during the study.
* Taking dietary supplements, prescriptions, or over the counter medication, other than a contraceptive (unless approved by OMSO & PI).
* Abnormal blood count during OMSO medical screening (For example: hemoglobin (Hb) outside of the typical normal values reported by LabCorp in accordance with OMSO (Normal [Hb] Males = 12.6-17.7 g/dL; Females = 11.1-15.9 g/dL) or hematocrit (Hct) outside of the normal ranges (Normal Hct Males = 37.5-51.0%; Females = 34.0-46.6%) levels, presence of abnormal blood chemicals (hemoglobin S or sickle cell traits).
* Any history of pulmonary, cardiovascular, or renal disease (unless approved by OMSO & PI).
* Uncontrolled asthma.
* Current or recent respiratory tract or sinus infections (< 2 weeks prior).
* History of heat stroke or orthostatic intolerance.
* Diagnosed and/or treated for fluid/electrolyte imbalance within the last 30 days.
* History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis.
* Scheduled MRI during testing.
* Allergies to adhesives (e.g., medical tape).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
End-exercise Core Temperature | Through study completion, an average of 8 weeks
  End-exercise core temperature during heat stress test
Resting Core Temperature | Through study completion, an average of 8 weeks
  Core Temperature at Rest during Heat Stress Test
End-exercise heart rate | Through study completion, an average of 8 weeks
  Heart rate at end of heat stress test
End-exercise Mean Weighted Skin Temperature | Through study completion, an average of 8 weeks
  Mean weighted Skin temperature at end of heat stress test

SECONDARY OUTCOMES:
Urine Specific Gravity | Through study completion, an average of 8 weeks
  Urine specific gravity prior to heat stress test

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT07099872/ICF_000.pdf